## ISOMETRIC CORE MUSCLE ENDURANCE IN HEALTHY ACTIVE AND NON-ACTIVE WORKING AGE POPULATIONS Hanna Holmberg, Lynne E Gaskell

28.05.2018

## ISOMETRIC CORE MUSCLE ENDURANCE IN HEALTHY ACTIVE AND NON-ACTIVE WORKING AGE POPULATIONS

## Hanna Holmberg, Lynne E Gaskell

This is the first study to investigate the core muscle endurance of different age groups and genders with all four endurance tests of the core.

Core endurance has been previously tested in literature with either isometric or dynamic tests. Strand et al. (1), however, claim that dynamic tests like sit-ups are more indicative of inner range muscle strength and power, and therefore, do not reflect the muscle endurance. Biering-Sorensen, McGill v-sit and side plank have been found to be the most reliable and safe in a myriad of different isometric core endurance tests (2–7). The reliability of v-sit has been found to be 0.66-0.73 (7–9), Biering-Sorensen 0.54-0.99 (5,7,9) right side plank (RSP) 0.74-0.78 and left side plank (LSP) 0.91-0.96 (7,8) in healthy adult populations with and without low back pain (LBP).

Core endurance may be affected by different factors. Correia et al. (10) found that core muscle activity of people who experience LBP is delayed, which may lead to further dysfunction and pain. It is unclear, though, if reduced core muscle endurance affects LBP experience or the risk of its' development.

Another possible factor influencing the core muscle endurance is age. However, the results in the older general population are contradicting (mean age values of 37–47.95) (11,12) due to possible influence of participants' lifestyle, work, and selected endurance tests. We are living in an aging society and further investigation should be carried out to reject or confirm this possible connection.

As a result of aging, a healthy person loses 1–2% of the muscle mass (13–15) and put on 0.45kg fat every year after reaching the age of 40 (16,17). An increase in BMI has been associated with reduced core muscle endurance (18-20). However, physical activity may reduce these changes and account for different results of previous studies.

The purpose of this study was to investigate a possible correlation between core muscle endurance and participants' age in healthy adult population. The secondary purpose was to identify other dependent variables influencing isometric core muscle endurance (e.g. low back pain, physical activity, gender, body mass index).

48 (35 females, 13 males) healthy adults (aged 21–66 years) will perform 4 isometric core muscle endurance tests- Biering-Sorensen, McGill V-sit, right and left side plank. All

participants will be divided into 2 age groups considering the physiological changes taking place during aging- <41 and >40.

Guidelines suggest that to maintain a healthy lifestyle, adults aged between 18 and 65 should do moderate-intensity aerobic physical activities for a minimum of 30 minutes, 5 times a week, or high-intensity aerobic activities 20 minutes, 3 times a week (21–24). Participants will also be divided based on the physical activity level- groups that meets national and international guidelines and a group that doesn't. A correlation between core endurance and age, gender, low back pain (LBP), physical activity level (PAL), and body mass index (BMI) is calculated using Pearson's correlation and Independent T-test on SPSS. It is a case control study, collecting both numerical and categorical data.

- 1. Strand SL, Hjelm J, Shoepe TC, Fajardo MA. Norms for an isometric muscle endurance test. Journal of Human Kinetics. 2014;40(1):93–102.
- 2. Champagne A, Descarreaux M, Lafond D. Comparison between elderly and young males' lumbopelvic extensor muscle endurance assessed during a clinical isometric back extension test. Journal of Manipulative and Physiological Therapeutics. 2009;32(7):521–6. Available from: http://dx.doi.org/10.1016/j.jmpt.2009.08.008
- 3. Dejanovic A, Balkovec C, McGill S. Head posture influences low back muscle endurance tests in 11-year-old children. Journal of Motor Behavior. 2015;47(3):226–31.
- 4. Demoulin C, Boyer M, Duchateau J, Grosdent S, Jidovtseff B, Crielaard JM, et al. Is the Sorensen test valid to assess muscle fatigue of the trunk extensor muscles? Journal of Back and Musculoskeletal Rehabilitation. 2016;29(1):31–40.
- 5. Moreau CE, Green BN, Johnson CD, Moreau SR. Isometric back extension endurance tests: A review of the literature. Journal of Manipulative and Physiological Therapeutics. 2001;24(2):110–22.
- 6. Musalem LL, Stankovic T, Glisic D, Cook GE, Beach TAC. Biomechanical and electromyographic comparisons of isometric trunk flexor endurance test postures: Prone plank versus V-sit. Journal of Applied Biomechanics. 2015;31(6):469–75.
- 7. Waldhelm A, Li L. Endurance tests are the most reliable core stability related measurements. Journal of Sport and Health Science. 2012;1(2):121–8.
- 8. Greene PF, Durall CJ, Kernozek TW. Intersession reliability and concurrent validity of isometric endurance tests for the lateral trunk muscles. Journal of Sport Rehabilitation. 2012;21(2):161–6.
- 9. Saeterbakken A. Muscle Activity, and the Association between core strength, core endurance and core stability. Journal of Novel Physiotherapy and Physical Rehabilitation. 2015;2(2):28–34.
- Correia JP, Oliveira R, Vaz JR, Silva L, Pezarat-Correia P. Trunk muscle activation, fatigue and low back pain in tennis players. Journal of Science and Medicine in Sport. 2016;19(4):311–6. Available from: <a href="http://dx.doi.org/10.1016/j.jsams.2015.04.002">http://dx.doi.org/10.1016/j.jsams.2015.04.002</a>
- 11. Del Pozo-Cruz B, Mocholi MH, Del Pozo-Cruz J, Parraca JA, Adsuar JC, Gusi N.

- Reliability and validity of lumbar and abdominal trunk muscle endurance tests in office workers with nonspecific subacute low back pain. Journal of Back and Musculoskeletal Rehabilitation. 2014;27(4):399–408.
- 12. Tekin Y, Ortancil O, Ankarali H, Basaran A, Sarikaya S, Ozdolap S. Biering-Sorensen test scores in coal miners. Joint Bone Spine. 2009;76(3):281–5. Available from: http://dx.doi.org/10.1016/j.jbspin.2008.08.008
- 13. Hughes VA, Frontera WR, Roubenoff R, Evans WJ, Fiatarone Singh MA. Longitudinal changes in body composition in older men and women: Role of body weight change and physical activity. American Journal of Clinical Nutrition. 2002;76(2):473–81.
- 14. Landi F, Cherubini A, Cesari M, Calvani R, Tosato M, Sisto A, Martone AM, Bernabei R, Marzetti E. Sarcopenia and frailty: From theoretical approach into clinical practice. European Geriatric Medicine. 2016;7(3):197–200. Available from: http://dx.doi.org/10.1016/j.eurger.2015.12.015
- 15. Perkisas S, De Cock A-M, Verhoeven V, Vandewoude M. Intramuscular adipose tissue and the functional components of sarcopenia in hospitalized geriatric patients. Geriatrics. 2017;2(1):11.
- 16. Forbes GB. Longitudinal changes in adult fat-free mass: Influence of body weight. American Journal of Clinical Nutrition. 1999;70(6):1025–31.
- 17. Kohrt WM, Bloomfield SA, Little KD, Nelson ME, Yingling VR. Physical activity and bone health position stand. Medicine and Science in Sports and Exercise. 2004;36(11):1985–96.
- 18. Mayer JM, Nuzzo JL, Chen R, Quillen WS, Verna JL, Miro R, et al. The impact of obesity on back and core muscular endurance in firefighters. Journal of Obesity. 2012;2012.
- 19. Kankaanpää M, Laaksonen D, Taimela S, Kokko SM, Airaksinen O, Hänninen O. Age, sex, and body mass index as determinants of back and hip extensor fatigue in the isometric Sorensen back endurance test. Archives of Physical Medicine and Rehabilitation. 1998;79(9):1069–75.
- 20. Ummunah JO, Ibikunle PO, Ezeakunne AC. Relationship between isometric endurance of back extensor muscles and selected anthropometric indices among some Nigerian undergraduates. Journal of Back and Musculoskeletal Rehabilitation. 2014;27(3):291–

- 21. Haskell WL, Lee IM, Pate RR, Powell KE, Blair SN, Franklin BA, et al. Physical activity and public health: Updated recommendation for adults from the American College of Sports Medicine and the American Heart Association. Medicine and Science in Sports and Exercise. 2007;39(8):1423–34.
- 22. Hupin D, Roche F, Gremeaux V, Chatard JC, Oriol M, Gaspoz JM, et al. Even a low-dose of moderate-to-vigorous physical activity reduces mortality by 22% in adults aged ≥60 years: A systematic review and meta-analysis. British Journal of Sports Medicine. 2015;49(19):1262–7.
- 23. Kahlmeier S, Wijnhoven TMA, Alpiger P, Schweizer C, Breda J, Martin BW. National physical activity recommendations: Systematic overview and analysis of the situation in European countries. BMC Public Health. 2015;15:133.
- Piercy KL, Troiano RP, Ballard RM, Carlson SA, Fulton JE, Galuska DA, George SM OR. The physical activity guidelines for Americans. JAMA Journal of the American Medical Association. 2018;320(19):2020–8.